CLINICAL TRIAL: NCT04623944
Title: A Phase 1 Study of NKX101, an Activating Chimeric Receptor Natural Killer Cell Therapy, in Subjects With Hematological Malignancies or Dysplasias
Brief Title: NKX101, Intravenous Allogeneic CAR NK Cells, in Adults With AML or MDS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nkarta, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKX101-101
Record Dates: First submitted 2020-09-25; First posted 2020-11-10 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Relapsed/Refractory AML; AML, Adult; MDS; Refractory Myelodysplastic Syndromes
Keywords: NKG2D; CAR; Allogeneic; Natural killer; ACR; NKX101; IL15; Interleukin 15; NK cell; Cell Therapy; Immunotherapy; Adoptive cell therapy; r/r AML; Off-the-shelf
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Cyclophosphamide; fludarabine; Cytarabine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NKX101 - CAR NK cell therapy (Experimental): All subjects in Part 1 will receive lymphodepletion with fludarabine/cyclophosphamide followed by 3 or 2 (Regimen A or B, respectively) weekly doses of NKX101.
  Subjects in Part 2 will receive lymphodepletion with either fludarabine/cyclophosphamide or fludarabine/cytarabine (ara-C), or if the optional arm is opened, lymphodepletion with fludarabine/cyclophosphamide and decitabine, followed by 3 weekly doses of NKX101.
  Part 2: unrelated off-the-shelf donor derived NKX101 will be used.
  Interventions: Biological: NKX101 - CAR NK cell therapy

INTERVENTIONS:
Biological: NKX101 - CAR NK cell therapy — NKX101 is an investigational allogeneic CAR NK product targeting NKG2D ligands on cancer cells. Part 2 will use the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of NKX101 as determined in Part 1.
  Other Names: Cyclophosphamide; Fludarabine; Cytarabine (ara-C); Decitabine

SUMMARY:
This is a single-arm, open-label, multi-center, Phase 1 study to determine safety and tolerability of an experimental therapy called NKX101 (allogeneic CAR NK cells targeting NKG2D ligands) in patients with relapsed/refractory AML or intermediate, high and very high risk relapsed/refractory MDS.

DETAILED DESCRIPTION:
This is a dose-finding study of NKX101 and will be conducted in 2 parts:

Part 1: dose finding with two dosing regimens, utilizing modified "3+3" enrollment schema.

Part 2: dose expansion to further evaluate safety and tolerability, cellular kinetics, pharmacodynamics and anti-tumor response in expansion cohorts of patients with either AML or MDS.

ELIGIBILITY:
Inclusion Criteria:

* General:

  * ECOG performance status ≤2
* Disease related:

  * For AML subjects:

    * Previously treated relapsed/refractory AML, including subjects with MRD+ disease
    * Received at most 3 lines of previous anti-leukemia therapy
    * For subjects with targetable fms-like tyrosine kinase 3 (FLT3)-mutated or isocitrate dehydrogenase (IDH)1/2 mutated disease, subjects must have received at least 1 prior respective targeted therapy and may receive up to 4 lines of prior therapy
    * White blood cell count of ≤25 × 10^9/L
    * For groups receiving NKX101 after lymphodepletion with fludarabine/cyclophosphamide +/- decitabine: Disease localized to the bone marrow, as evidenced by ≤ 5% peripheral blasts and no evidence of extramedullary disease
    * For groups receiving NKX101 after lymphodepletion with fludarabine/ cyclophosphamide +/- decitabine, group receiving NKX101 after lymphodepletion with fludarabine/ara-C: Additional subjects with specifically high-risk genetic mutations may be enrolled. High risk genetic mutation per ELN 2022 should be evaluated as per local assay and discussed with the Sponsor prior to study entry
    * For groups receiving NKX101 after lymphodepletion with fludarabine/cyclophosphamide +/- decitabine, group receiving NKX101 after lymphodepletion with fludarabine/ara-C: Additional subjects who have relapsed following HCT may be enrolled.
  * For MDS subjects:

    * Intermediate-, high-, or very high-risk MDS
    * Previously treated relapsed/refractory MDS
    * Received at least 1 and at most 3 lines of previous standard anti-MDS therapy
    * For groups receiving NKX101 after lymphodepletion with fludarabine/ cyclophosphamide +/- decitabine: Additional subjects with specifically high-risk disease may be enrolled. High-risk genetic mutation should be evaluated as per local assay
    * For group receiving lymphodepletion with fludarabine/cyclophosphamide +/- decitabine and NKX101: Additional subjects who have relapsed following HCT may be enrolled.
* Adequate Organ Function
* Platelet count ≥30,000/uL (platelet transfusions acceptable)
* Other:

  * Signed informed consent
  * Agree to use an effective barrier method of birth control

Exclusion Criteria:

* Disease related:

  * Acute promyelocytic leukemia with t(15;17) (q22;q12); or abnormal promyelocytic leukemia/retinoic acid receptor alpha (APML-RARA) and AML arising from chronic myelomonocytic leukemia (CMML)
  * Evidence of leukemic meningitis or known active central nervous system disease
  * Peripheral leukocytosis with ≥ 20,000 blasts/μL or other evidence of rapidly progressive disease that would preclude subject from completing at least 1 cycle of treatment
  * Use of any anti-AML/MDS chemotherapeutic or targeted small molecule drug within protocol specified window prior to the first dose of NKX101
  * Presence of residual non-hematologic toxicity from prior therapies that has not resolved to ≤ Grade 1
  * Any hematopoietic cell transplantation within 16 weeks
* Other comorbid conditions and concomitant medications prohibited as per study protocol
* Other:

  * Pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2039-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 30 days after last dose of NKX101
  Incidence, nature, and severity of treatment related adverse events will be evaluated. An adverse event is any unfavorable and unintended sign including clinically significant abnormal laboratory findings, symptom or disease.
Response rate to NKX101 (for Part 2) | 28 days from first dose of NKX101
  Responses will be assessed per modified ELN criteria and will include complete and partial remission with and without varying degrees of hematologic recovery

SECONDARY OUTCOMES:
Assessment of NKX101 half-life | 28 days from first dose of NKX101
  Time required for 50% reduction from maximum amount of circulating NKX101
NKX101 duration of persistence | Followed up to 2 years after last dose of NKX101
  Testing NKX101 in peripheral blood every 3 months after dosing to determine persistence
Evaluation of host immune response against NKX101 | Followed up to 2 years after last dose of NKX101
  Serum samples will be measured for antibodies against NKX101
Response rate to NKX101 | Primary assessment: 28 days after first dose of NKX101 followed up to 2 years after last dose of NKX101
  Time-to-first response, time-to-best response, duration of response, transfusion independent rate, bridge-to-transplant rate, event-free survival, progression-free survival (PFS), overall survival (OS) (for all subjects), and hematologic improvement rates (for subjects with myelodysplastic syndrome [MDS])

CONTACTS AND LOCATIONS:
Overall Officials: David Shook, MD, Study Director — Nkarta, Inc.
Locations (8):
- United States (8):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - The Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Sarah Cannon at TriStar Bone Marrow Transplant Center, Nashville, Tennessee
  - MD Anderson Cancer Center, University of Texas, Houston, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No